CLINICAL TRIAL: NCT03652246
Title: Evaluation of the Diagnostic Contribution of High-throughput Exome Sequencing for Patients With Convulsive Encephalopathy of Unknown Etiology: Pilot Study to Improve Genetic Counselling
Acronym: SHD-EE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Masurel-Thevenon AOI 2013
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Epileptic Encephalopathy of Unindentified Genetic Origin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital epileptic encephalopathies (EE) are predominantly genetic in origin. Their diagnosis is hampered by the large number of genes involved and their low recurrence. Genetic study in routine diagnosis is limited by the existing techniques and the development costs. The routine diagnostic implementation of high throughput sequencing pushes these limits. High throughput exome sequencing (ES) showed superior diagnostic performance in all diagnostic settings studied.

This pilot study is dedicated to evaluating the diagnostic performance of high throughput ES in EE, with an implementation and analysis strategy allowing for a direct transfer to routine diagnostics. This novel approach should improve the diagnostic rate while reducing the diagnostic cost per patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epileptic encephalopathy, defined by the clinical association of epilepsy and a significant delay in acquisition
* Family case with recurrence in siblings, suggesting autosomal recessive transmission or X-linked inheritance (with or without parental consanguinity), or sporadic case resulting from inbreeding.
* Lack of etiologic orientation based on clinical examination.
* Normal routine diagnostic genetic examinations including a metabolic check-up, array CGH analysis.
* Brain imaging which does not suggest an acquired cause.

Exclusion Criteria:

* Unavailable parental samples
* Diagnostic orientation from one of the tests mentioned above
* Brain imaging suggesting anoxia sequelae

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient in consultation
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of diagnoses performed with high throughput ES | Through study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France